CLINICAL TRIAL: NCT04731584
Title: Systemic Inflammation During Recanalization of Cerebral Arterial Occlusion
Acronym: CONVASC-I
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1080
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Systemic Infection
MeSH Terms: conditions — Stroke; Toxemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AVC: Patients hospitalized for TM after a proximal ischemic stroke of the middle cerebral artery and whose reperfusion is satisfactory (TICI 2b, 2c and 3). Additional blood sample will be taken during usual treatment the day of the stroke.
  Interventions: Biological: Blood sample
- Control: Population of control patients, consisting of patients admitted on an outpatient basis for a diagnostic cerebral arteriography.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Patients from 2 groups will undergo blood sample (during a blood sample for there care) and inflammation parameters will be measure the day of the stroke

SUMMARY:
Strokes management, secondary to proximal arterial occlusion, by endovascular thrombectomy (TM) is now well established. The immuno-inflammatory events of reperfusion after TM are discussed. Systemic inflammation is a major factor suggested to explain the limited recovery of the ischemic parenchyma. Understanding these phenomena is necessary before developing an immunomodulatory strategy.

ELIGIBILITY:
GROUP "AVC" :

Inclusion Criteria:

* Adults patient (s)
* Ischemic stroke by occlusion of a middle cerebral artery (proximal portion M1)
* Initial diagnostic MRI infusion
* TM with complete reperfusion (TICI 2b, 2c or 3)
* TM performed under local anesthesia +/- anxiolysis, or sedation including propofol
* mRS prior to stroke <2
* Barthel index <90
* Included in the HIBISCUS cohort
* Patient who was informed and did not object to participating in the study OR included through the emergency procedure then collection of his non-objection or that of his trusted person as soon as possible

Exclusion Criteria:

* NIHSS awareness score> or = 2
* Haemorrhagic complication before thrombectomy
* Pregnant woman
* Multiple vascular occlusions
* Occlusions of posterior or anterior cerebral territories other than M1
* Protected major
* TM performed under general anesthesia
* Other vital failure than neurological failure

GROUP "CONTROL" :

Inclusion Criteria:

* Adults patient (s)
* mRS <2
* Barthel index <90
* Requiring diagnostic arteriography for routine check-up of a cerebrovascular malformation
* Patient who was informed and did not object to participating in the study

Exclusion Criteria:

* NIHSS awareness score> or = 2
* Pregnant woman
* Protected major
* Exam performed under general anesthesia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for TM after a proximal ischemic stroke of the middle cerebral artery and whose reperfusion is satisfactory (TICI 2b, 2c and 3).
  Population of control patients, consisting of patients admitted on an outpatient basis for diagnostic cerebral arteriography.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Inflammation parameters description | 1 day
  Inflammatory parameters such as CRP, IL-6, IL-10, HLA-DR, TNF-alpha, polymorphonuclear chemotaxis, CD-4, T-lymphocytes will be measure in blood sample

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service d'Anesthésie Réanimation Hôpital - Neurologique/Groupement Est, Bron
  - Service de Neurologie vasculaire - Hôpital Neurologique/Groupement Est, Bron
  - Service de Neuroradiologie interventionnelle - Hôpital Neurologique/Groupement Est, Bron
  - Service d'Anesthésie Réanimation - Hôpital Edouard Herriot/Groupement Centre, Lyon

IPD SHARING:
Plan to Share IPD: No